CLINICAL TRIAL: NCT00482781
Title: Prolonged Apnea and Prolonged Bradycardia Following DTaP Immunization in Preterm Infants: A Randomized Multicenter Study
Brief Title: DTaP and Apnea/Bradycardia in Preterm Infants
Acronym: PIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American SIDS Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PIA-09012000
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-06

CONDITIONS: Prolonged Apnea; Prolonged Bradycardia
Keywords: Apnea; Bradycardia; Preterm Infant; Immunization; DTaP
MeSH Terms: conditions — Apnea; Bradycardia; Premature Birth | interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Infanrix
Biological: Pediatrix

SUMMARY:
The purpose of this study is to examine the relationship between receipt of DTaP and the occurrence of prolonged episodes of apnea and bradycardia in preterm infants, while employing a random control study design and an objective assessment of cardiorespiratory events.

DETAILED DESCRIPTION:
The American Academy of Pediatrics (AAP) recommends the immunization of preterm infants at two months chronological age with the diphtheria-tetanus-acellular pertussis (DTaP) vaccine, regardless of birth weight and gestational age. However, several investigators, employing historical controls and subjective observations, have reported an increased incidence in prolonged apnea and bradycardia in preterm infants following immunization. Consequently, many primary care providers do not adhere to recommended AAP guidelines. The purpose of this study is to reexamine the relationship between receipt of DTaP and the occurrence of prolonged episodes of apnea and bradycardia in preterm infants, while employing a random control study design and an objective assessment of cardiorespiratory events.

Ten participating hospitals will enroll infants < 37 completed weeks gestational age into the study when they are 56-60 days chronological age. Infants are randomly assigned into one of two groups: One group receives DTaP immunization and the control group does not (until study is completed). Physiological event recording monitors are used continuously during the next 2 days to document the incidence of prolonged apnea (respiratory pause of ≥20 sec in duration or >15 sec in duration if associated with bradycardia for ≥5 sec) and prolonged bradycardia (heart rate <80 bpm that lasted ≥10 sec) in all infants. The presence and number of episodes during the 48-hour period will be compared between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Born at a gestational age < 37 weeks.
* Still in the hospital at time of study.
* Between 56 - 60 days chronological age.

Exclusion Criteria:

* Had active infections, were critically ill, or had unstable vital signs.
* Requiring assisted ventilation or tracheostomy during the study.

Ages: 56 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 191 (Actual)
Dates: Start 2000-09; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Bedside recording of apnea and bradycardia with events verified by 2 independent scorers who were blinded to the study phase and immunization status of the subject. | Six days (Three 48-hour periods).

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Carbone, MD, Principal Investigator — Valley Hospital, Ridgewood, NJ; Betty McEntire, PhD, Study Director — American SIDS Institute
Locations (10):
- United States (10):
  - Wellstar Cobb Hospital, Austell, Georgia
  - Kennestone Hospital, Marietta, Georgia
  - St. Peters Univ. Hospital, Belle Mead, New Jersey
  - Brooklyn Hospital, Brooklyn, New York
  - St. Joseph's Hospital Health Ctr., Syracuse, New York
  - Toledo Children's Hospital, Toledo, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - The Children's Home of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital, Greenville, South Carolina

REFERENCES:
- [Derived] Carbone T, McEntire B, Kissin D, Kelly D, Steinschneider A, Violaris K, Karamchandani N. Absence of an increase in cardiorespiratory events after diphtheria-tetanus-acellular pertussis immunization in preterm infants: a randomized, multicenter study. Pediatrics. 2008 May;121(5):e1085-90. doi: 10.1542/peds.2007-2059. PMID 18450851